CLINICAL TRIAL: NCT01069718
Title: Evaluating the Effect of Patterned Oral Somatosensory Entrainment Stimulation Using the NTrainer on Oral Feeding Performance in Infants With Feeding Dysfunction
Brief Title: Evaluating Patterned Oral Somatosensory Entrainment Stimulation Using the NTrainer on Oral Feeding Performance
Status: Completed | Type: Observational
Sponsor: KC BioMediX, Inc (Industry)
Responsible Party: Thomas Young, MD, WakeMed Faculty Physician
Other Study IDs: WakeMEd Study 751
Record Dates: First submitted 2010-02-15; First posted 2010-02-17 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2010-02

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Clinical Group: In the Clinical group bottle feedings will be attempted by the bedside nurses, using techniques suggested in the feeding plan. The Infant Feeding Specialist will observe at least one feeding per day to assure that the feeding plan is being adhered to. If, in the judgment of the person feeding the infant, the infant is unable to complete the bottle feeding, the remaining volume will be given via an indwelling gavage tube. During all gavage feedings, both total and partial, infants will be offered a pacifier to suck on.
- NTrainer Group: In the NTrainer group, three feedings per day will be given via gavage tube while the infant is receiving NTrainer stimulation. The stimulation will be done by alternating 3 minute epochs of NTrainer stimulation with 3 minutes of sucking on a regular pacifier, up to a total time of 30 minutes.
  Every other day, 15 minutes prior to a feeding that is not one of the study sessions, each infant's suck strength and coordination will be measured using the NTrainer device in its "NeoSuck RT" Assessment mode.
  On the day after the study intervention period is completed each infant will be assessed by an investigator unaware of the infant's study group assignment.

SUMMARY:
This is a research study to determine if an experimental device called the NTrainer can improve oral feeding skills more quickly and more effectively than traditional methods in infants who are at high risk of feeding dysfunction and delayed hospital discharge.

DETAILED DESCRIPTION:
One day prior to starting the study treatment, sucking strength and coordination will be measured on all enrolled infants using the NTrainer device in its "NeoSuck RT" assessment mode (See Appendix A). They will also be clinically assessed by an Infant Feeding Specialist using clinical assessment tools including the NOMAS and EFS (see Appendix B). After the assessment a feeding plan will be developed for use by the infant's bedside nurses. This feeding plan will include but not be limited to the use of techniques such as oromotor stimulation, side-lying, pacing, and slow flow nipples. After the clinical and NeoSuck assessments, infants will be randomized to receive either "Clinical" or "NTrainer" intervention. The intervention period will be 10 days.

For study intervention feedings, the infant will undergo a brief exam of physiologic state, using the Oral Feeding Readiness Assessment portion of the EFS. If the infant is determined to be ready to feed (s)he infant will be cradled in a supportive inclined posture, swaddled, with limbs positioned at midline, and background/overhead lighting dimmed in the area. The infant will remain connected to the usual ICN monitors at all times for observation of respiration, heartbeat and oxygen saturation.

In the Clinical group bottle feedings will be attempted by the bedside nurses, using techniques suggested in the feeding plan. The Infant Feeding Specialist will observe at least one feeding per day to assure that the feeding plan is being adhered to. If, in the judgment of the person feeding the infant, the infant is unable to complete the bottle feeding, the remaining volume will be given via an indwelling gavage tube. During all gavage feedings, both total and partial, infants will be offered a pacifier to suck on.

In the NTrainer group, three feedings per day will be given via gavage tube while the infant is receiving NTrainer stimulation. The stimulation will be done by alternating 3 minute epochs of NTrainer stimulation with 3 minutes of sucking on a regular pacifier, up to a total time of 30 minutes. Bottle feedings will be attempted at the other daily feedings by the bedside nurse using techniques suggested by the feeding plan. If the infant is unable to complete the bottle feeding, the remaining volume will be given via an indwelling gavage tube. During all gavage feedings, both total and partial, infants will be offered a pacifier to suck on.

Every other day, 15 minutes prior to a feeding that is not one of the study sessions, each infant's suck strength and coordination will be measured using the NTrainer device in its "NeoSuck RT" Assessment mode.

If the infant is able to successfully bottle feed the full prescribed volume for 5 of 8 feedings per 24 hours, the study intervention will end.

On the day after the study intervention period is completed each infant will be assessed by an investigator unaware of the infant's study group assignment. The assessment will include (1) a 3-minute measurement of sucking strength and coordination using "NeoSuck RT", and (2) two observational checklists (NOMAS and EFS) used to score infant feeding behaviors. The amount of oral feeding as a percentage of daily feeding volume will be recorded, as well as the number of feeding-associated apnea/bradycardia/oxygen desaturation events in the preceding 24 hours.

The NTrainer recordings will be interpreted by researchers at the University of Kansas, but each baby's medical information will be kept confidential. The NTrainer study results will not become part WakeMed records. Each baby's study records will be available through the Neonatology division of WakeMed Faculty Physicians.

ELIGIBILITY:
Inclusion Criteria:

* 34 weeks postmenstrual age, medically stable enough to attempt bottle feedings
* Born at 28 completed weeks of gestation or less and are still on oxygen at 34 weeks postmenstrual age, or (2) have had intestinal surgery, or (3) have had recurrent episodes of feeding intolerance, or (4) have a significant intracranial hemorrhage or periventricular leukomalacia.

Exclusion Criteria:

* Infants will be excluded if their mothers plan to exclusively breastfeed their infant after discharge home.

Ages: 34 Weeks to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants born prematurely may suffer multiple adverse events in the Intensive Care Nursery, and these experiences may negatively impact normal developmental processes of immature cardiorespiratory, gastrointestinal and central nervous systems. As a result, many infants have at least transient difficulties learning to successfully manage oral feedings. Oral feeding difficulties in the ICN may prolong the time to discharge, cause significant parental anxiety, and persist throughout infancy. Indeed, as many as 40% of patients followed in feeding disorder clinics are former preterm infants.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2008-03; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Postmenstrual age at the time of full oral feedings | At the time of full oral feedings
Postmenstrual age at the time of hospital discharge | At discharge

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Young, MD, Principal Investigator — Wake Med Faculty Physician
Locations (1):
- WakeMed, Raleigh, North Carolina, United States

REFERENCES:
- [Background] Barlow SM, Finan DS, Lee J, Chu S. Synthetic orocutaneous stimulation entrains preterm infants with feeding difficulties to suck. J Perinatol. 2008 Aug;28(8):541-8. doi: 10.1038/jp.2008.57. Epub 2008 Jun 12. PMID 18548084